CLINICAL TRIAL: NCT01280344
Title: Phase II Double-Blind Placebo-Controlled Dose Finding Study to Evaluate Safety/Efficacy of Ipamorelin Compared to Placebo for Recovery of Gastrointestinal Function in Patients Following Small or Large Bowel Resection w/Primary Anastomosis
Brief Title: Safety and Efficacy of Ipamorelin Compared to Placebo for the Recovery of Gastrointestinal Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Therapeutics (U.S.), Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT-IPAM-202
Record Dates: First submitted 2011-01-13; First posted 2011-01-20 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Gastrointestinal Dysmotility
MeSH Terms: interventions — Saline Solution; Injections; ipamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.03 mg/kg BID (Experimental): Ipamorelin 0.03 mg/kg, BID (2 investigational drug infusions and 1 placebo infusion)
  Interventions: Drug: Ipamorelin
- 0.06 mg/kg BID (Experimental): Ipamorelin 0.06 mg/kg, BID (2 investigational drug infusions and 1 placebo infusion)
  Interventions: Drug: Ipamorelin
- 0.06 mg/kg TID (Experimental): Ipamorelin 0.06 mg/kg, TID (3 investigational drug infusions)
  Interventions: Drug: Ipamorelin
- Placebo (Placebo Comparator): Matching placebo, TID (3 placebo infusions)
  Interventions: Drug: Saline Solution for Injection

INTERVENTIONS:
Drug: Saline Solution for Injection — Intravenous (IV)
  Arms: Placebo
Drug: Ipamorelin — Intravenous (IV)
  Arms: 0.03 mg/kg BID; 0.06 mg/kg BID; 0.06 mg/kg TID

SUMMARY:
Post-operative administration of ipamorelin is expected to reduce time to recovery of Gastrointestinal (GI) function in patients who have undergone partial small and/or large bowel resection.

ELIGIBILITY:
Inclusion Criteria:

* Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form
* Males or females, 18 to 85 years of age inclusive at the time of study screening
* American Society of Anesthesiologists (ASA) Class I-III
* Have undergone a scheduled small and/or large open partial bowel resection based on a documented incision size greater than or equal to (≥) 10 cm with primary anastomosis
* Females must not be pregnant as confirmed by a serum pregnancy test at screening and by a urine pregnancy test on the day of surgery
* Body weight must be between 40-150 kilograms (kg)

Exclusion Criteria:

* Any procedure which requires a diverting stoma
* Primary anastomosis not performed at the time of surgery
* Epidural or intrathecal anesthesia
* Significant liver disease (ALT and/or total bilirubin > 2-fold upper limits of normal) or kidney disease (serum creatinine > 2.5 mg/dL) at screening
* History of irritable bowel syndrome
* Patients with a history of Crohn's disease or ulcerative colitis (UC) who have had multiple GI-related surgeries (Note: surgery naïve Crohn's or UC patients may be included)
* History of colonic volvulus
* History of gastroesophageal surgery, gastrectomy, gastric bypass, total colectomy, short bowel syndrome, or multiple complex abdominal surgeries performed by an open procedure (uncomplicated cesarean section and appendectomy would not be considered complex)
* Patients who have received prior abdominal radiation and/or pelvic radiation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Recovery of Gastrointestinal (GI) Function | Up to 10 days
  To assess the efficacy of three repeated dose levels of ipamorelin vs. placebo

SECONDARY OUTCOMES:
Ancillary GI Functions | Up to 10 days or until hospital discharge
  To investigate the effect of ipamorelin on ancillary efficacy measures of GI function and recovery
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | 14 day outpatient follow-up visit
  To investigate the safety and tolerability of ipamorelin laboratory and clinical parameters, incidence of adverse events, until hospital discharge, 14-day outpatient follow-up visit, or until resolution of adverse events

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Florence, Alabama
  - Sheffield, Alabama
  - Fountain Valley, California
  - Glendale, California
  - Laguna Hills, California
  - Los Angeles, California
  - Orange, California
  - San Francisco, California
  - Aurora, Colorado
  - Aventura, Florida
  - Inverness, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Highland Park, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Springfield, Massachusetts
  - Flint, Michigan
  - Royal Oak, Michigan
  - Troy, Michigan
  - Jackson, Mississippi
  - St Louis, Missouri
  - Stony Brook, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Nassau Bay, Texas
  - Burlington, Vermont
  - Bellevue, Washington
  - Milwaukee, Wisconsin